CLINICAL TRIAL: NCT02497261
Title: Early Life Origins of the Food Allergy Epidemic: Predictors of Persistent Peanut Allergy at Age 5 Years
Brief Title: Predictors of Persistent Peanut Allergy at Age 5 Years
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: University of British Columbia (Other); The Hospital for Sick Children (Other); McGill University (Other)
Responsible Party: Principal Investigator, Elinor Simons, Dr. Elinor Simons, Assistant Professor, University of Manitoba
Other Study IDs: B2015:052
Record Dates: First submitted 2015-06-04; First posted 2015-07-14 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Allergy to Peanut
Keywords: Food Allergy; Peanut; Sensitization; Child; Double-blind placebo-controlled challenge; Prospective cohort
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for immunological markers of peanut allergy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Avoiding and possibly allergic to peanut: Challenge Group: Children with positive skin prick testing to peanut who are avoiding peanut will undergo a double-blind placebo-controlled peanut challenge (gold standard for peanut allergy diagnosis) if their allergy evaluation suggests that they have a good chance of not being allergic to peanut. Children who pass the challenge are not allergic to peanut. Children who react during the challenge are allergic to peanut and will continue to avoid peanut.
  Interventions: Procedure: Double-blind placebo-controlled peanut challenge
- Not allergic to peanut: Comparison Group: Children with positive skin prick testing to peanut who are eating and tolerating peanut are not clinically allergic to peanut and may continue eating peanut.

INTERVENTIONS:
Procedure: Double-blind placebo-controlled peanut challenge — Children who are avoiding peanut will be gradually introduced to smoothies containing and not containing peanut, to see if they are able to tolerate eating peanut. This challenge does not change a child's ability to tolerate peanut, but will determine which children avoiding peanut are allergic to peanut and which children are not allergic and may begin eating peanut.
  Other Names: Tiny 1st peanut dose & scheduled doses increased by 1/2-log; No drugs or devices
  Groups: Avoiding and possibly allergic to peanut

SUMMARY:
The purpose of this study is to determine if avoidance of peanut by children with positive allergy testing to peanut in the first 5 years of life increases the likelihood of developing a persistent peanut allergy by age 5 years. To answer this question, the investigators need to determine which children with positive allergy testing to peanut have reactions after eating peanut (allergic to peanut) and which are able to tolerate eating peanut (not allergic).

The investigators plan to conduct double-blind placebo-controlled peanut challenges (gold standard for peanut allergy diagnosis) for CHILD study (http://www.canadianchildstudy.ca) participants who had positive skin prick testing to peanut at ages 1, 3 or 5 years (in other words, children who are sensitized to peanut, but may or may not be allergic to peanut) and who are avoiding peanut without ever having had a reaction or whose history suggests that they may have outgrown a known peanut allergy. These challenges will not change a child's ability to tolerate peanut, but will determine if children who are avoiding peanut are allergic to peanut (and need to continue avoiding peanut) or clinically tolerant to peanut (and may continue to eat peanut after passing the challenge).

DETAILED DESCRIPTION:
Introduction:

Food allergy has reached epidemic levels in Canada and peanut allergy is the most prevalent and one of the more persistent food allergies among Canadian children and adults. Avoidance or later introduction of peanut has been proposed as a possible cause of the increased rates of peanut sensitization and allergy. Although delaying the introduction of peanut into children's diets is no longer recommended, many parents continue to worry about introducing peanut and some will not introduce peanut into their child's diet without a negative skin prick test to peanut. However, some children who have never had a reaction to peanut can eat and tolerate peanut despite being sensitized (having a positive skin prick test) to peanut.

The purpose of this study is to determine if avoidance of peanut by children with positive skin prick testing to peanut in the first 5 years of life increases the likelihood of developing a persistent peanut allergy by age 5 years. To answer this question, the investigators need to determine which children with positive skin prick testing to peanut have reactions after eating peanut (allergic to peanut) and which are able to tolerate eating peanut (not allergic).

Specific Objectives:

1. To conduct double-blind placebo-controlled peanut challenges among 5-year-old children who are sensitized to and avoiding peanut, to determine if they are allergic to peanut (and need to continue avoiding peanut) or clinically tolerant to peanut (and may continue to eat peanut after passing the challenge)
2. To determine the relative risk of developing peanut allergy among peanut-sensitized children who have been eating versus avoiding peanut.

Challenge Procedure:

Double-blind placebo-controlled food challenges are the gold standard clinical practice for diagnosis of food allergies, and involve the child undergoing separate challenges to the food and to a placebo so that the child, parents, and physicians and nurses administering the challenge are masked regarding which challenge is to the food and which is to the placebo. All children will undergo challenges to both peanut and placebo, in a randomized order. These challenges will not change a child's ability to tolerate peanut, but will determine if children who are avoiding peanut are allergic to peanut (and need to continue avoiding peanut) or clinically tolerant to peanut (and may continue to eat peanut after passing the challenge).

The challenges will be conducted in clinical units set up for food challenges, by a research nurse and a pediatric allergist with expertise and experience in managing food allergies and oral food challenges. Each child will undergo a challenge to peanut on one day and a challenge to placebo on another day. The peanut will be concealed in a vehicle, such as a shake or smoothie. One of the challenges will contain peanut and the concealing vehicle and the other challenge will contain only the vehicle. The challenge foods will be prepared by a team member who is not otherwise involved in the challenges. A study worker not involved in the challenges will also be in charge of randomizing the two challenges to peanut or placebo and of decoding the challenge food identity after both challenges are completed. The children, their families, the research nurse and the pediatric allergist will not know whether the challenge food contains the peanut or the placebo until both challenges have been completed. This procedure helps to distinguish symptoms that occur due to anxiety (equally likely to occur in both the peanut and placebo challenges) and those that are a reaction to peanut (occur only during the peanut challenge).

Children who do not develop any symptoms of anaphylaxis (e.g. hives, swelling, trouble breathing, vomiting, abdominal pain or changes in their level of consciousness) during the challenge or the 2-hour observation period after the challenge will have passed the challenge and will be considered clinically tolerant; they will be encouraged to continue eating peanut at home at least once per week. Children who develop any of these symptoms during the challenge containing peanut will be considered allergic, especially if symptoms did not occur during the challenge containing only the vehicle.

ELIGIBILITY:
Challenge Inclusion Criteria:

CHILD study participants will be eligible for challenge if they

1. Have completed their 5-year-old CHILD Study visit
2. Are or have been sensitized to peanut i.e. have had a positive skin prick test (wheal diameter at least 2 mm greater than the negative control) and/or allergen-specific IgE level (>0.35 kU/L) to peanut at their 1-, 3- and/or 5-year-old CHILD study visit
3. Are not eating peanut. Children who eat less than 8-10 g of peanut per month or who eat only foods that 'may contain' traces of peanut will still be eligible for inclusion.

Challenge Exclusion Criteria:

CHILD study participants will be ineligible for challenge if

1. They have never had a positive skin prick test or allergen-specific IgE level to peanut
2. They are eating 8-10 g of peanut at least once per month, despite having had a positive skin prick test or allergen-specific IgE level to peanut
3. Their family has declined to participate
4. They have a peanut skin prick test wheal size >8mm and/or a peanut-specific IgE >15 kU/L and a history suggestive of an IgE-mediated allergic reaction to peanut.
5. They have a history of anaphylaxis to peanut or a challenge-proven diagnosis of peanut allergy within the past 1-2 years.
6. They have uncontrolled asthma or any other contraindication to performing a DBPC food challenge on the day of challenge. These children may be rescheduled if their asthma control improves.

Blood Draw Inclusion Criteria:

CHILD study participants will be eligible for blood draw if they

1. Have completed their 5-year-old CHILD Study visit
2. Are or have been sensitized to peanut i.e. have had a positive skin prick test (wheal diameter at least 2 mm greater than the negative control) and/or allergen-specific IgE level (>0.35 kU/L) to peanut at their 1-, 3- and/or 5-year-old CHILD study visit

Blood Draw Exclusion Criteria:

CHILD study participants will be ineligible for blood draw if

1. They have never had a positive skin prick test or allergen-specific IgE level to peanut
2. Their family has declined to participate

Immunological analyses of the blood samples are underway now that the 2 sites participating in this portion of the study (University of Manitoba and University of British Columbia) have completed their challenges. Challenges were halted in the spring.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited from among the participants of the Canadian Healthy Infant Longitudinal Development (CHILD) Study (http://www.canadianchildstudy.ca) who have completed their 5-year-old study visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical tolerance to peanut (passing a peanut challenge and eating peanut regularly) | Age 5 years
  Clinical tolerance to peanut (passing a peanut challenge and eating peanut regularly)

CONTACTS AND LOCATIONS:
Overall Officials: Elinor Simons, MD PhD MSc, Principal Investigator — Section of Allergy, Department of Pediatrics & Child Health, University of Manitoba

IPD SHARING:
Plan to Share IPD: Undecided